CLINICAL TRIAL: NCT07063823
Title: A First-in-human Study to Evaluate the Safety and Tolerability of HB-2121 as a Diagnostic for Celiac Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nielsen Fernandez-Becker (Other)
Collaborators: Stanford's Innovative Medicines Accelerator (Unknown)
Responsible Party: Sponsor-Investigator, Nielsen Fernandez-Becker, Clinical Professor, Medicine - Gastroenterology & Hepatology, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-80209
Record Dates: First submitted 2025-06-16; First posted 2025-07-14 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-06

CONDITIONS: Celiac Disease; Healthy
Keywords: Celiac Disease; HB-2121; Healthy Volunteers; Gluten Intolerance
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- 50 mg HB-2121 in Healthy Volunteers (Experimental): Participants in this arm will receive a one-time dose of 50 mg of HB-2121.
  Interventions: Drug: HB-2121
- 150 mg HB-2121 in Healthy Volunteers (Experimental): Participants in this arm will receive a one-time dose of 150 mg of HB-2121.
  Interventions: Drug: HB-2121
- 250 mg HB-2121 in Healthy Volunteers (Experimental): Participants in this arm will receive a one-time dose of 250 mg of HB-2121.
  Interventions: Drug: HB-2121
- 50 mg HB-2121 in Participants with Celiac Disease (Experimental): Participants in this arm will receive a one-time dose of 50 mg of HB-2121.
  Interventions: Drug: HB-2121
- 150 mg HB-2121 in Participants with Celiac Disease (Experimental): Participants in this arm will receive a one-time dose of 150 mg of HB-2121.
  Interventions: Drug: HB-2121
- 250 mg HB-2121 in Participants with Celiac Disease (Experimental): Participants in this arm will receive a one-time dose of 250 mg of HB-2121.
  Interventions: Drug: HB-2121

INTERVENTIONS:
Drug: HB-2121 — HB-2121 taken once orally.

SUMMARY:
The goal of this clinical trial is to learn about the safety of a single dose of HB-2121 in adults. It will also look at how the body processes the drug. The main questions it aims to answer are:

* What side effects do participants have after receiving HB-2121?
* How much HB-2121 is in the blood over time?

Researchers will follow participants for 30 days after receiving HB-2121 to understand how the drug behaves in the body and how safe it is.

Participants will:

* Receive one oral dose of HB-2121
* Attend 4 in-person clinic visits for checkups, lab tests, and monitoring
* Complete 2 remote visits that include safety lab assessments
* Fill out a short daily questionnaire for 7 days about symptoms and health status

ELIGIBILITY:
General Inclusion Criteria (applies to all participants):

* Aged 18 years and older
* Body Mass Index (BMI) between 18 and 45 kg/m2
* Overall good health, as determined by medical history and a physical exam
* No use of an investigational drug in the past 12 weeks
* Able and willing to follow study procedures and provide written informed consent
* If of childbearing potential, participants must agree to use highly effective birth control during the study period. The same applies to male participants with partners of childbearing potential

Additional Inclusion Criteria for Healthy Volunteers:

* No diagnosis of celiac disease
* No first-degree relatives (parent, sibling, child) with celiac disease
* Able to eat gluten-containing foods without adverse effects
* No history of autoimmune gastrointestinal disorders such as Crohn's disease, ulcerative colitis, or eosinophilic enteritis

Additional Inclusion Criteria for Participants with Celiac Disease:

* Biopsy-confirmed diagnosis of celiac disease
* No history of eosinophilic enteritis, autoimmune gastrointestinal disorders such as Crohn's disease or inflammatory bowel disease

Exclusion Criteria (applies to all participants):

* Pregnant, breastfeeding, or planning to become pregnant during the study period
* History of chemotherapy or pelvic radiation
* History of congenital long QT syndrome or prolonged QTcF interval
* Known HIV infection, or positive test for hepatitis B or C, or other clinically significant chronic liver disease
* Current use of immunosuppressant medications
* Known allergy or sensitivity to any ingredients in the study drug
* Active cancer or history of cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-08-26 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of adverse events during the study window | From dosing through 30 days post-dose
  Adverse events (AEs) will be recorded and assessed for severity using the Common Terminology Criteria for Adverse Events (CTCAE) v5.0.

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) of HB-2121 | Pre-dose, and at 15, 30, 60, 120, 180, 240, and 360 minutes, and 1 day after dosing.
  Blood samples will be collected at specified time points to determine the peak plasma concentration (Cmax) of HB-2121 following administration.
Time to Peak Plasma Concentration (Tmax) of HB-2121 | Pre-dose, and at 15, 30, 60, 120, 180, 240, and 360 minutes, and 1 day after dosing.
  Time to reach the maximum plasma concentration (Tmax) of HB-2121 will be determined from blood sample data collected at specified time points.
Area Under the Plasma Concentration-Time Curve (AUC) for HB-2121 | Pre-dose, and at 15, 30, 60, 120, 180, 240, and 360 minutes, and 1 day after dosing.
  The area under the plasma concentration versus time curve (AUC) for HB-2121 will be calculated using plasma concentration data from collected blood samples.

OTHER OUTCOMES:
Frequency and identity of HB-2121 positive cells in the blood of healthy subjects and patients with celiac disease | 60, 120, 180, 240, and 360 minutes, and 1 day after dosing
  Blood samples will be collected after dosing, and peripheral blood mononuclear cells (PBMCs) will be analyzed using flow cytometry to determine the percentage of HB-2121+ cells among CD14+CD11c+ populations, with and without β7-integrin expression.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States